CLINICAL TRIAL: NCT04314778
Title: Using Patient Centered Data and Behavioral Economics to Improve Mobility and Reduce Readmissions After Major Abdominal Surgery for Cancer
Brief Title: FITBIT Study on Mobility and Readmissions After Radical Cystectomy
Acronym: FITBIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Daniel Lee, MD, MS, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 833829
Record Dates: First submitted 2020-01-09; First posted 2020-03-19 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention arm will have a postoperative daily step goal that increases from baseline by 500 steps each day.
  Interventions: Behavioral: social incentive-based gamification
- Control (No Intervention): Participants in the control group will have data collected passively via Fitbit.

INTERVENTIONS:
Behavioral: social incentive-based gamification — At the beginning of each week, starting from postoperative day 3, the participant receives 70 points (10 points for each day that week). If the participant does not meet their daily step goal, they lose 10 points from their balance. This leverages loss aversion, which has been demonstrated to motivate behavior change more effectively with losses than gains. At the end of each week if the participant has at least 40 points, they will move up a level (levels from lowest to highest: blue, bronze, silver, gold, platinum). If not, the participant will drop a level. All participants begin at the silver level. Each week, participants get a fresh set of 70 points. Participants will receive daily feedback for the step counts, and weekly feedback for their levels. Participants in the intervention arm will be asked to identify a family member or friend to be their support sponsor. A weekly report will be sent to this person with the participant's performance (points and level).
  Arms: Intervention

SUMMARY:
This is a two-arm randomized, controlled trial during the postoperative period after major abdominal surgery for cancer, including for example radical cystectomy, nephrectomy, colectomy, comparing a control group that uses a wearable device to track physical activity to an intervention group that uses the same wearable devices and receives a supportive social incentive-based gamification intervention to adhere to a step goal program.

DETAILED DESCRIPTION:
We will conduct a two-arm randomized, controlled trial during the postoperative period after a radical cystectomy for bladder cancer, comparing a control group that uses a wearable device to track physical activity to an intervention group that uses the same wearable devices and receives a supportive social incentive-based gamification intervention to adhere to a step goal program. Patients will be enrolled after being diagnosed with bladder cancer and scheduled to undergo a radical cystectomy. The median length of stay after a radical cystectomy is 8 days, with 90% being discharged within two weeks. Postoperatively, the baseline step count will be averaged by taking the steps taken during the first two days outside of the intensive care unit. There will be two postoperative phases: Phase I will be while the patient is hospitalized postoperatively. Phase II will be when the patient is discharged for three months.

5.2 Study

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* diagnosis of cancer undergoing definitive surgical treatment

Exclusion Criteria:

* Inability to provide consent
* does not have daily access to a smartphone compatible with the wearable device and not willing to use a device that the investigators can provide them
* any other medical conditions that would prohibit participation in a physical activity program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lee, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 64 participants gave informed consent but 3 participants declined to complete required pre-randomization surveys. These participants were not assigned to intervention or control groups and were excluded from the study.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 30 | 31
Completed | 25 | 28
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 64 patients gave informed consent but only 61 completed run-in and were randomized.
  years | 65.3 (10.2) | 67 (12.4) | 66.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 21 | 25 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 25 | 25 | 50
  Black, non-Hispanic | 4 | 4 | 8
  Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Daily Step Count From the Baseline Step Count During Two Days After the Surgery to the Hospital Discharge
Description: Change in mean daily step count
Time Frame: From baseline step count after a two-day run-in period after the surgery to the time of hospital discharge postoperatively. As the time to discharge was variable, this time period was up to 60 days after surgery
Population: Only 23 participants had recorded step count data of more than two days while in the hospital. This clinical trial was performed during the height of the COVID-19 pandemic when research staff and hospital staff were not allowed in the hospital or on University campuses, making follow up in the hospital difficult while patients were recovering from a major surgery
Measure: Mean (95% Confidence Interval); unit: mean change in daily steps
Arm/Group | Intervention | Control
Number analyzed (Participants) | 8 | 15
mean change in daily steps | 1087 [652 to 1521] | 995 [185 to 1806]

2. Secondary Outcome: Change in Mean Daily Step Count From the Postoperative Baseline to 3 Months After Discharge From the Hospital
Description: Change in mean daily step count
Time Frame: From the postoperative baseline step count during 2 day run-in to 3 months after discharge from the hospital. This time was up to 3 months after discharge
Measure: Mean (Standard Deviation); unit: mean change in daily steps
Groups:
- Intervention: gamification with support partner
- Control: Control
Arm/Group | Intervention | Control
Number analyzed (Participants) | 25 | 28
mean change in daily steps | 5674 (3681) | 4660 (3063)

3. Other Pre Specified Outcome: Rate of Placement to Skilled Nursing Facility After Hospital Discharge
Description: Rate of placement to skilled nursing facility postoperatively
Time Frame: 13 weeks after hospital discharge
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Rate of 90 Day Hospital Readmission After Hospital Discharge
Description: Rate of 90 day hospital readmission
Time Frame: 90 days after hospital discharge
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Rate of Postoperative Complications
Description: Rate of complications after the surgery
Time Frame: Immediately after the surgery to 3 months postoperatively
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Rate of Postoperative Delirium
Description: Rate of delirium after the surgery
Time Frame: Immediately after the surgery to 3 months postoperatively
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the study period of 6 months.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 0/30 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT04314778/Prot_SAP_000.pdf